CLINICAL TRIAL: NCT01769911
Title: AUTOLOGOUS TRANSPLANTATION AND STEM CELL BASED-GENE THERAPY FOR THE TREATMENT OF HIV-ASSOCIATED LYMPHOMA
Brief Title: Genetically Modified Peripheral Blood Stem Cell Transplant in Treating Patients With HIV-Associated Non-Hodgkin or Hodgkin Lymphoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2583.00; NCI-2012-03168 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH)
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; AIDS-related Diffuse Large Cell Lymphoma; AIDS-related Diffuse Mixed Cell Lymphoma; AIDS-related Diffuse Small Cleaved Cell Lymphoma; AIDS-related Immunoblastic Large Cell Lymphoma; AIDS-related Lymphoblastic Lymphoma; AIDS-related Peripheral/Systemic Lymphoma; AIDS-related Small Noncleaved Cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; HIV-associated Hodgkin Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage I AIDS-related Lymphoma; Stage II AIDS-related Lymphoma; Stage III AIDS-related Lymphoma; Stage IV AIDS-related Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Lymphoma, AIDS-Related; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Carmustine; Cytarabine; Melphalan; Etoposide; O(6)-benzylguanine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (gene modified peripheral blood cell transplant) (Experimental): CONDITIONING: Patients receive carmustine IV over 3 hours on day -7, cytarabine IV over 2 hours BID and etoposide IV over 2 hours BID on days -6 to -3, and melphalan IV over 30 minutes on day -2.
  TRANSPLANTATION: Patients receive an autologous PBSC infusion and/or infusion of autologous transduced hematopoietic cells on day 0.
  Beginning 28-120 days later, patients eligible for in vivo selection after detection of gene-marked cells receive O6-benzylguanine IV over 1 hour and carmustine IV over 3 hours on days 14, 28, and then monthly until completion of therapy. Patients achieving > 10% gene marking and CD4 count of >= 500 cells/uL receive up to 2 courses of structured treatment interruption without undergoing in vivo selection.
  Interventions: Drug: carmustine; Drug: cytarabine; Drug: melphalan; Drug: etoposide; Drug: O6-benzylguanine; Procedure: autologous hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: carmustine — Given IV
  Other Names: BCNU; BiCNU; bis-chloronitrosourea
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: O6-benzylguanine — Given IV
  Other Names: BG
Procedure: autologous hematopoietic stem cell transplantation — Undergo transduced and/or non-transduced transplant
Procedure: peripheral blood stem cell transplantation — Undergo transduced and/or non-transduced transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies genetically modified peripheral blood stem cell transplant in treating patients with HIV-associated non-Hodgkin or Hodgkin lymphoma. Giving chemotherapy before a peripheral stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. After treatment, stem cells are collected from the patient's blood and stored. More chemotherapy or radiation therapy is then given to prepare the bone marrow for the stem cell transplant. Laboratory-treated stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and radiation therapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and feasibility of infusing gene-modified, human immunodeficiency virus (HIV)-protected hematopoietic stem cells (HSC) after high-dose chemotherapy for treatment of acquired immunodeficiency syndrome (AIDS)-related lymphoma.

II. To determine the dose of carmustine (BCNU) in combination with O^6-benzylguanine (O6BG) that results in selection in vivo of gene-modified HIV-resistant cells.

III. To estimate the effect of HIV infection on the presence of HIV-resistant blood cells as measured by genetic marking for vector sequences before and after antiviral treatment interruption.

SECONDARY OBJECTIVES:

I. Evaluate the molecular and clonal composition of gene-modified cells after hematopoietic cell transplant (HCT).

II. Evaluate the molecular and clonal composition of gene-modified cells after O6BG/BCNU.

III. Determine the correlation of the level of O6-methylguanine- methyltransferase (MGMT) (P140K) marking with toxicity and response.

IV. Characterize the toxicity associated with in vivo selection. V. Determine the efficacy of the procedure for treatment of lymphoma: defined as time to disease progression, progression-free survival, treatment-related mortality, time to neutrophil and platelet recovery, and incidence of infections.

TERTIARY OBJECTIVES:

I. Effect of procedure on the latent HIV reservoir. II. Effect of procedure on HIV-specific immune reconstitution.

OUTLINE:

CONDITIONING: Patients receive carmustine intravenously (IV) over 3 hours on day -7, cytarabine IV over 2 hours twice daily (BID) and etoposide IV over 2 hours BID on days -6 to -3, and melphalan IV over 30 minutes on day -2.

TRANSPLANTATION: Patients receive an autologous PBSC infusion and/or infusion of autologous transduced hematopoietic cells on day 0.

Beginning 28-120 days later, patients eligible for in vivo selection after detection of gene-marked cells receive O6-benzylguanine IV over 1 hour and carmustine IV over 3 hours on days 14, 28, and then monthly until completion of therapy. Patients achieving > 10% gene marking and CD4 count of >= 500 cells/uL receive up to 2 courses of structured treatment interruption without undergoing in vivo selection.

After completion of study treatment, patients are followed up periodically for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive
* Antiretroviral treatment for at least one month, defined as a multi-drug regimen (excluding azacitidine [AZT])
* HIV plasma viral load has decreased by 1.5 logs or viral load < 5000 copies/ml
* Non-Hodgkin or Hodgkin lymphoma without active central nervous system (CNS) involvement associated with poor prognosis with medical therapy alone or for which autologous peripheral blood stem cell (PBSC) transplant is indicated:

  * Hodgkin's lymphoma beyond first remission; first partial remission; induction failure with subsequent response to salvage therapy
  * Non-Hodgkin's Lymphoma beyond first remission: first partial remission; induction failure with subsequent response to salvage therapy
  * Chemotherapy responsive disease
* Karnofsky performance score >= 70%
* Subjects must agree to use effective contraception from enrollment through completion of the study
* Female subjects: if of child bearing potential, must have negative serum or urine pregnancy test within 7 days of treatment
* Subjects must be on a prophylactic regimen for Pneumocystis carinii pneumonia, or agree to begin such treatment, if the cluster of differentiation (CD)4 counts are =< 200
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Serum creatinine > 2 times upper limit of normal
* Serum bilirubin greater than 3 times the upper limits of normal, unless determined to be a result of the primary hematologic malignancy or attributed to Gilbert's syndrome
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 3 times the upper limits of normal, unless determined to be a result of the primary hematologic malignancy or attributed to Gilbert's syndrome
* Forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1) or diffusion capacity of the lung of carbon monoxide (DLCO) parameters < 60% predicted (corrected for hemoglobin)
* Left ventricular ejection fraction (LVEF) < 50% or coronary artery disease requiring treatment
* Active infection requiring systemic antibiotic therapy with antibacterial, antifungal, or antiviral agents (excluding HIV)
* Patients who are hepatitis C virus (HCV) antibody positive or hepatitis B virus (HBV) surface antigen positive must be free of clinical evidence of cirrhosis that would otherwise make them ineligible for HCT, as determined by the Principal Investigator (P.I.) in consultation with the Gastrointestinal Service; patients with HBV and ongoing evidence of viral replication may require therapy prior to receiving high-dose chemotherapy
* Positive serology for Toxoplasma gondii AND requiring treatment or with evidence of active infection
* Malignancy other than lymphoma, unless 1) in complete remission and more than 5 years from last treatment), or 2) cervical/anal squamous cell carcinoma in situ or 3) superficial basal cell and squamous cell cancers of the skin
* History of HIV-associated encephalopathy; dementia of any kind; seizures in the past 12 months; any perceived inability to directly provide informed consent (Note: Consent may not be obtained by means of a legal guardian)
* A medical history of noncompliance with highly active anti-retroviral therapy (HAART) or medical therapy

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Safety of infusion of gene-modified cells, measured by grade 3 or greater toxicities related to infusion of gene-modified cells using the Common Toxicity Criteria version 4.0(CTCv.4) | Up to day 180
Safety of O6BG/BCNU in vivo selection, defined as less than 25% of patients developing grade 3 or greater non-hematopoietic toxicity or grade 4 CTCv.4 hematopoietic toxicity | Up to day 180
Safety of structured treatment interruption defined as no decline in CD4 count by more than 25%, no HIV RNA more than 10,000 copies/mL; and no elevation of immune activation markers | During the 12 weeks without HAART
Efficacy of gene transduction, defined as collection of more than 4.5 x 10^6 CD34+ cells/kg cells for genetic modification and evidence of gene-marked cells before HSC infusion | Up to 3 months
Efficacy of infusion of gene-modified cells, defined as engraftment of at least1% gene-modified cells | Up to 3 months
Efficacy of O6BG/BCNU in vivo selection, defined as selection of gene-modified cells to a level at least 10% of peripheral blood cells | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ann Woolfrey, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States